CLINICAL TRIAL: NCT05275621
Title: Virtual Reality for Vascular Access: a Multicenter Feasibility Study
Brief Title: Virtual Reality as a Substitute to Pharmacological Sedation During PICC Placement in Pediatric Patients
Acronym: ViVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Marco Gemma, Director of Anesthesia and Intensive Care Unit, ASST Fatebenefratelli Sacco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/ST/291
Record Dates: First submitted 2022-02-14; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Procedural Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects requiring PICC (Experimental): Subjects requiring a PICC. Positioning is first tried under Virtual Reality distraction. If failure (movements or discomfort) standard procedural sedation is applied. No kind of physical restraint is allowed.
  Interventions: Device: Virtual Reality; Procedure: PICC positioning

INTERVENTIONS:
Device: Virtual Reality — A Virtual Reality game is provided through a headset. Subjects play in a virtual environment. Positioning of the headset occurs before starting the procedure and is maintained throughout the procedure. The headset used will be "Oculus Rift 2 by Facebook Tech. ltd.". The software is designed specifically for the purpose by Softcare Studios. The "game" played is called "Drums".
Procedure: PICC positioning — A PICC is inserted under ultrasound guidance through a modified Seldinger technique in a deep vein of the upper arm. The skin is infiltrated with 0.5-1ml 2% lidocaine before dilation of the skin. Tip guidance and positioning is achieved through intracavitary ECG.

SUMMARY:
In pediatric patients Peripherally Inserted Central Catheters (PICC) insertion requires pharmacological sedation provided by an anesthesiologist, which poses a certain degree of risks. In enrolled subjects, PICC insertion is tried without drug sedation, using an immersive virtual reality experience as a distraction technique. If the subjects is not able to keep still or if pain levels are too high, the virtual reality attempt is stopped and standard drug sedation is provided by a pediatric anesthesiologist.

Aim of study is to evaluate the feasibility of the PICC insertion procedure using the virtual reality distraction technique. The investigators hypothesize that this could avoid the need for drug sedation, reducing sedation-related risks and costs and reduce anxiety and pain related to the procedure.

DETAILED DESCRIPTION:
A PICC is a central intravenous catheter inserted through a peripheral vein of the upper arm. In pediatric subjects, the insertion usually requires pharmacological sedation because of the anxiety and the pain experienced by the children during the procedure. Sedation inevitably poses a certain risk, particularly of airway obstruction, respiratory drive reduction en hemodynamic instability. Finally, costs are sensibly higher when sedation is required, since, besides the need for drugs and devices (e.g. for monitoring and airway management), an experienced pediatric anesthesiologist and a nurse are needed for providing sedation.

The investigators hypothesize that the application of virtual reality to children undergoing PICC placement, could avoid the need for drug sedation. This would result in a reduction in anxiety and pain related to the procedure and a potential reduction in costs. Moreover any possible adverse event related to pharmacological sedation would be avoided.

The material used for providing the virtual reality experience consist of a commercially available virtual reality headset (Oculus Quest 2 by Facebook Technologies ltd) and a dedicated software called "TOMMI" (developed by Softcare Studios Srl). Subjects find themselves in a virtual environment where they can play different games. The game which was chosen is called "drums", optimized for enhanced sensorimotor engagement and distraction from acute sensations such as pain. In this game subjects see three different drums they can beat with a "magic wand" they can control by moving the handheld controller. Geometric shapes in different colors fall from above indicating which drum to beat and at which time.

This game was chosen for several reasons: it can be played for sufficient time without getting excessively boring or tiring (the procedure usually lasts about half an hour); it can be easily played both by younger and older children; it does not require wide movements either of the head or of the upper limb holding the controller, and the opposite upper limb isn't involved in any way. Thus, distracting or even dangerous movements of the subject can be avoided, ensuring the successful completion of the procedure.

Subjects will be enrolled by the investigators in each participating center according to the inclusion and exclusion criteria. To participate informed consent has to be acquired in written form from both the caregivers and, if able to do so, also by the subjects.

Before the procedure multiple variables will be recorded to draw a baseline of each enrolled subject. These will include age, sex, BMI, previous experiences of sedation and of venipuncture and a psychological and behavioral profile using a self-administered questionnaire for caregivers (Child Behaviour Checklist - Achenbach ASEBA).

At the start of the procedure the Investigators will explain to the subject the use of the Virtual Reality viewer and will help him in positioning it. Patients will be monitored with continuous ECG and SpO2. All PICC placements will be carried out by trained and experienced implanter, in a dedicated room and under full barrier precautions. A pediatric anesthesiologist will always be available on site.

While arranging the sterile field, and at least for five minutes, the implanter will let the patient get fully immersed in the virtual environment. Meanwhile, the implanter will check that the child has correctly understood how to play the game.

In each patient, the site of insertion will be chosen after proper echographic evaluation of the vascular anatomy following the RaPeVA protocol as recommended by the Italian Vascular Access Society (IVAS). Entry site will be chosen in the middle third of the upper arm or in the "green zone" after the Zone Insertion Method™ by Robert Dawson. Venipuncture will be performed under ultrasound guidance and the catheter will be placed using a modified Seldinger technique over a tearaway introducer. Before introducing the dilator, the provider will inject the area with a local anesthetic and performed a small skin incision with a scalpel. Tip guidance and location was achieved through continuous intracavitary ECG.

Standard procedural sedation will be provided for those who won't tolerate the procedure using only the Virtual Reality immersion. No kind of active or passive restraint will be enforced during the whole procedure, the patients will be required to hold still for the whole time just by themselves.

Data will be analyzed with the R software in its latest version - Copyright (C) 2021 The R Foundation for Statistical Computing Platform: R Core Team (2021). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL https://www.R-project.org/.

Continuous data will be reported as mean and standard deviation, categorical as number (percentage).

The investigators consider the accomplishment of the PICC placement procedure as the primary endpoint of our study (a dichotomous N/Y variable).

The procedure with the virtual reality is expected to be successful in the majority of all cases. Hence, in calculating the sample size (without finite population correction), the investigators consider an expected proportion of accomplishment of 0.95 with a precision (half width of the 95 percent confidence interval) of 0.04. This yields a sample size of 120 patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 7 and 14 years old
* Indication for Vascular Access Device placement with the need for sedation
* Signed informed consent form by the subject's caregivers (commonly both parents)

Exclusion Criteria:

* Inability to fill in the rating scales
* Inability to experience Virtual Reality with TOMMI (e.g., eye diseases)
* Presence of disease that produces complete immobility
* Refusal to sign informed consent

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change in baseline Pain assessed by the Wong-Baker FACES Scale | Baseline and Five minutes after the procedure has been completed
  The Wong-Baker FACES Scale is a validated scale used to assess the experienced pain in subjects from three years of age. It consists of six different faces: the first represents no pain at all and is described by the words "No Hurt" and the last one represents a pain score of "10 out of 10" on a numeric rating scale, and indicates "hurts worst."
Change in baseline Anxiety assessed by a numeric rating scale | Baseline and Five minutes after the procedure has been completed
  Anxiety is assessed through a numeric rating scale ranging from zero representing no anxiety at all, up to ten representing the worst anxiety level.

SECONDARY OUTCOMES:
Duration of the procedure | During the procedure
  time for catheter positioning is measured
Subject's satisfaction | through study completion, an average of three months
  Subject's satisfaction is measured through a numeric rate scale from 0 to 10 with 0 indicating extreme discomfort and 10 indicating absolute satisfaction.
Staff satisfaction | After study completion, expected six months
  Staff satisfaction on the procedure is evaluated through a numeric rate scale from 0, indicating not satisfied at all, to 10, very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Gemma, MD, Principal Investigator — ASST Fatebenefratelli Sacco
Locations (6):
- Italy (6):
  - Spedali Civili di Brescia, Brescia, BS
  - Ospedale Pediatrico Istituto Gianna Gaslini, Genova, GE
  - Ospedale dei Bambini "Vittore Buzzi", Milan, MI
  - Fatebenefratelli Hospital, Milan, MI
  - AORN Pausilipon, Napoli
  - Regina Margherita Hospital, Torino

IPD SHARING:
Plan to Share IPD: No